CLINICAL TRIAL: NCT05987384
Title: The Role of Fatty Acids in Vaccine Efficacy: A Randomized Controlled Clinical Trial
Brief Title: The Role of Fatty Acids in Vaccine Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tsinghua University (Other)
Responsible Party: Principal Investigator, Ai Zhao, Assistant Professor, Tsinghua University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 20220081
Record Dates: First submitted 2023-06-08; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Rabies Vaccination Reaction
Keywords: Rabies Vaccination; Arachidonic acid; efficacy
MeSH Terms: interventions — Arachidonic Acid; Sunflower Oil; Rabies Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): Sunflower oil capsules
  Interventions: Dietary Supplement: Sunflower oil; Biological: Rabies Vaccine (Vero Cell) for Human Use
- D3 ARA group (Experimental): ARA capsules
  Interventions: Dietary Supplement: Arachidonic acid; Biological: Rabies Vaccine (Vero Cell) for Human Use
- D6 ARA group (Experimental): Sunflower oil capsules and ARA capsules
  Interventions: Dietary Supplement: Arachidonic acid; Dietary Supplement: Sunflower oil; Biological: Rabies Vaccine (Vero Cell) for Human Use

INTERVENTIONS:
Dietary Supplement: Arachidonic acid — D3 ARA group will receive ARA capsules from the third day of the study. D6 ARA group will receive ARA capsules from the sixth day of the study
  Arms: D3 ARA group; D6 ARA group
Dietary Supplement: Sunflower oil — The placebo group and D6 ARA group will receive sunflower oil capsules from the third day of the study. D6 ARA group will stop receiving sunflower oil capsules from the fifth day of the study.
  Arms: D6 ARA group; Placebo group
Biological: Rabies Vaccine (Vero Cell) for Human Use — Every participant will receive three doses of rabies vaccination.

SUMMARY:
This study intends to use a randomized controlled trial design to vaccinate all participants against rabies and perform ARA interventions during vaccination to test the efficacy, safety, and intestinal flora of each group after immunization.

DETAILED DESCRIPTION:
Rabies is an acute zoonotic infectious disease caused by central nervous system invasion by rabies virus. At present, there is still a lack of effective treatment, and once clinical symptoms appear, it is almost 100% fatal. Rabies vaccination within 24 hours of exposure may reduce the incidence of rabies. Pre-exposure prophylaxis is also effective, and the current recommended pre-exposure vaccination program in China is 0 days, 7th day, 21st days.

The health of the human body is inseparable from various nutrients. There are studies suggesting that arachidonic acid(ARA) has an immunomodulatory effect, but there is limited evidence for its effect on vaccines. Therefore, this study will explore the effects of nutritional supplements on the effectiveness of rabies vaccination.

ELIGIBILITY:
Inclusion Criteria:

* 1）18-45 years old;
* 2）BMI 18.5-24.9 kg/m2;
* 3）Have not received rabies vaccination.

Exclusion Criteria:

* 1) Those who have severe disorders of abnormal lipid metabolism;
* 2) Those who have used lipid-lowering drugs, weight loss drugs, and insulin drugs in the past three months;
* 3) Those who have received other vaccines in the past three months;
* 4) Those who have used probiotics or prebiotics in the past three months;
* 5) Those who have used steroids and immunosuppressants, other hormonal drugs in the past year;
* 6) Those with immunodeficiency diseases;
* 7) Those with a history of severe vaccine allergies;
* 8) Those who have disorders of liver and kidney metabolism;
* 9) Those who have had fever, cold, severe diarrhea and other diseases in the past month.
* 10) Smokers in the last year.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Changes of rabies virus antibody titers | Day 6, 13, 16, 19, 26 of the study
  specific antibody titers
Changes of neutralizing antibody titers | Day 6, 13, 16, 19, 26 of the study
  To test the ability of binding to rabies virus

SECONDARY OUTCOMES:
serum blood fatty acid profiles | Day 6, 13, 16，19 of the study
  to test the change of fatty acid profiles after intervention
C-reactive protein | Day 6, 13, 16 and 19 of the study
  to test the potential C-reactive protein changes triggered by ARA supplementation
Routine analysis of intestinal flora: alpha diversity | Day 3 and day 19 of the study
  The alpha diversity of microbiota in feces samples will be examined to explore the potential gut-immune response caused by intervention.
Routine analysis of intestinal flora: beta diversity | Day 3 and day 19 of the study
  The beta diversity of microbiota in feces samples will be examined to explore the potential gut-immune response caused by the intervention.
Routine analysis of intestinal flora: species abundance histogram | Day 3 and day 19 of the study
  The species abundance histogram of microbiota in feces samples will be examined to explore the potential gut-immune response caused by the intervention.
Routine analysis of intestinal flora: Lefse | Day 3 and day 19 of the study
  The Lefse of microbiota in feces samples will be conducted to explore the potential gut-immune response caused by the intervention.
Routine analysis of intestinal flora: PLS-DA | Day 3 and day 19 of the study
  The PLS-DA of microbiota in feces samples will be conducted to explore the potential gut-immune response caused by the intervention.
Routine analysis of intestinal flora: KEGG pathway | Day 3 and day 19 of the study
  The KEGG pathway microbiota in feces samples will be analyzed to explore the potential gut-immune response caused by the intervention.
Routine analysis of intestinal flora: differential KO expression | Day 3 and day 19 of the study
  The differential KO expression microbiota in feces samples will be analyzed to explore the potential gut-immune response caused by the intervention.
Macrogenomic sequencing difference of intestinal flora | Day 3 and day 19 of the study
  The macrogenomic sequencing analysis of microbiota in feces samples will be conducted to explore the potential gut-immune response caused by the intervention.
Fecal fatty acid content | Day 3 and day 19 of the study
  The fatty acid content in feces samples will be examined to explore the change of fatty acid intake caused by the intervention.

OTHER OUTCOMES:
Adverse events by ARA | Day 3 to day 30 of the trial.
  To examine the safety of using ARA, including allergy, gastrointestinal discomfort and others.
Serum triglyceride levels | Days 3 and day 19 of the study.
  To examine the changes of blood lipids in blood after intervention and evaluate the intervention safety. The spacific measurements include: Triglycerides (TG), high-density lipoprotein cholesterol (HDL-CHO), low-density lipoprotein cholesterol (LDL-C), and total cholesterol (TC).
Blood count: red blood cells | tested on day 3 and day 19 of the trial.
  To evaluate the intervention safety.
Blood count: white blood cells | tested on day 3 and day 19 of the trial.
  To evaluate the intervention safety.
Blood count: hemoglobin | tested on day 3 and day 19 of the trial.
  To evaluate the intervention safety.
Blood count: hematocrit | tested on day 3 and day 19 of the trial.
  To evaluate the intervention safety.
Blood count: platelets | tested on day 3 and day 19 of the trial.
  To evaluate the intervention safety.
Anxiety | tested on day 13 of the trial.
  Evaluated with General Anxiety Disorder-7 items. The scores are between 0 to 21, higher scores mean a worse outcome.
Depression | tested on day 13 of the trial.
  Evaluated with Patient Health Questionaire-9 items. The scores are between 0 to 27, higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ai Zhao, Doctor, Study Chair — Tsinghua University
Locations (1):
- Tsinghua University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen T, Welburn SC, Sun L, Yang GJ. Progress towards dog-mediated rabies elimination in PR China: a scoping review. Infect Dis Poverty. 2023 Apr 6;12(1):30. doi: 10.1186/s40249-023-01082-3. PMID 37024944

DOCUMENTS (2):
  • Study Protocol (2023-05-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT05987384/Prot_000.pdf
  • Informed Consent Form (2023-05-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT05987384/ICF_001.pdf